CLINICAL TRIAL: NCT04335760
Title: Is There a Relationship Between Fear of Activity and Functional Capacity in Patients With Coronary Artery Disease? - A Multi-Center Study From Turkey
Brief Title: Fear of Activity and Functional Capacity in Patients With Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Tuğba Atan (Other)
Responsible Party: Sponsor-Investigator, Tuğba Atan, MD, Physiatrist (Department of Physical Medicine and Rehabilitation), Hitit University
Organization: Hitit University (Other)
Other Study IDs: 25901600/7587, 27.11.2013
Record Dates: First submitted 2020-04-03; First posted 2020-04-06 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Coronary Artery Disease: Fear of activity scale in CAD (FactCAD) was used to assess fear of activity and exercise in subjects with CAD. FactCAD is a novel scale developed specifically for patients with heart disease. Mean time to complete this self-administered scale is 4-7 minutes. The final score of the questionnaire ranges between 0 and 84. High scores indicate higher levels of fear regarding activity or exercise.
  Functional capacity was assessed by 6MWT and exercise test. The 6MWT was performed to all participants according to the American Thoracic Society guidelines in a 30-m corridor10. The subjects were asked to walk as long distance as they could within 6 minutes. The 6MWT distance was recorded in meters.
  Exercise test was performed using modified Bruce protocol on treadmill in institutions where technical equipment and experience was available.
  Interventions: Combination Product: Modified Bruce protocol on treadmill
- healthy subjects: Fear of activity scale in CAD (FactCAD) was used to assess fear of activity and exercise in subjects with CAD. FactCAD is a novel scale developed specifically for patients with heart disease. Mean time to complete this self-administered scale is 4-7 minutes. The final score of the questionnaire ranges between 0 and 84. High scores indicate higher levels of fear regarding activity or exercise.
  Functional capacity was assessed by 6MWT and exercise test. The 6MWT was performed to all participants according to the American Thoracic Society guidelines in a 30-m corridor10. The subjects were asked to walk as long distance as they could within 6 minutes. The 6MWT distance was recorded in meters.
  Exercise test was performed using modified Bruce protocol on treadmill in institutions where technical equipment and experience was available.
  Interventions: Combination Product: Modified Bruce protocol on treadmill

INTERVENTIONS:
Combination Product: Modified Bruce protocol on treadmill — Fear of activity scale in CAD (FactCAD) was used to assess fear of activity and exercise in subjects with CAD. FactCAD is a novel scale developed specifically for patients with heart disease. Mean time to complete this self-administered scale is 4-7 minutes. The final score of the questionnaire ranges between 0 and 84. High scores indicate higher levels of fear regarding activity or exercise.
  Functional capacity was assessed by 6MWT and exercise test. The 6MWT was performed to all participants according to the American Thoracic Society guidelines in a 30-m corridor10. The subjects were asked to walk as long distance as they could within 6 minutes. The 6MWT distance was recorded in meters.
  Exercise test was performed using modified Bruce protocol on treadmill in institutions where technical equipment and experience was available.

SUMMARY:
To identify whether coronary artery disease (CAD) patients have fear of activity, and to assess the relationship between fear of activity and exercise capacity in CAD patients.

DETAILED DESCRIPTION:
Cardiac rehabilitation (CR) is a well-known way of secondary prevention in heart diseases. CR is shown to be effective in reducing cardiovascular morbidity and mortality. CR also enhances exercise capacity and quality of life, promotes healthy and active lifestyle and reduces psychosocial stress and depressive symptoms in coronary artery disease (CAD). Exercise is one of the most important component of CR. The positive prognostic effect of the exercise on cardiovascular disease is mediated by mechanisms such as reducing numerous risk factors, enhancing endothelial function, declining arterial inflammation and stiffness, improving diastolic function, remodeling of left ventricle, and stabilization of electrical activity. Each 1 MET increase in functional capacity is known to improve survival by 12 %. Exercise capacity is a more powerful predictor of mortality among men than other established risk factors for cardiovascular disease.

The prevalence of fear of activity in CAD, heart failure and female patients have been studied by several researchers reporting variable results. It ranges from 70% in acute hospitalized CAD patients to 20% in chronic patients in community. Muscle endurance, steps per day measured by pedometer, IPAQ were found to be lower in patients with high level of fear of activity.They did not measure exercise capacity objectively. Research investigating the effect of fear of activity on exercise capacity in patients with CAD is lacking.

The aim of this study is to identify whether coronary artery disease (CAD) patients have fear of activity, and to assess the relationship between fear of activity and exercise capacity in CAD patients. The hypothesis of this study were that CAD patients would have lower exercise capacity than healthy subjects and CAD patients with higher fear of activity would have lower exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* History of diagnosis of CAD and/or cardiac event in the past 1-60 months
* Being medically stable
* Cognitive and physical ability to complete the required tests.

Exclusion Criteria:

* Patients with recent cardiac event sooner than 1 month
* Musculoskeletal/neurologic problems imparing ambulation or current hospitalization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population consisted of 196 patients with CAD (144 men, 52 women) and 113 healthy subjects (73 men, 40 women).
Sampling Method: Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Fear of activity scale in CAD (FactCAD) | baseline
  Fear of activity scale in CAD (FactCAD) was used to assess fear of activity and exercise in subjects with CAD. FactCAD is a novel scale developed specifically for patients with heart disease. Mean time to complete this self-administered scale is 4-7 minutes. The final score of the questionnaire ranges between 0 and 84. High scores indicate higher levels of fear regarding activity or exercise.
Functional capacity (6MWT) | baseline
  Functional exercise capacity was assessed by distance walked in 6 minutes (6MWT). The patient was asked to walk as long as possible for 6 minutes on a 30 meters of marked and flat ground, at a self selected speed. 6MWT is a submaximal exercise test and can be used to assess treatment response.
Exercise test (Modified Bruce protocol) | baseline
  Modified Bruce protocol on treadmill was used in institutions where technical equipment and experience was available.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Medicine and Rehabilitation, Gaziler Physical Therapy and Rehabilitation Education and Research Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Multi-Center Study From Turkey — https://pubmed.ncbi.nlm.nih.gov/31562874/?from_term=tu%C4%9Fba+atan&from_pos=4